CLINICAL TRIAL: NCT04211324
Title: Acute Salivary Flow Rate Response to Transcutaneous Electrical Nerve Stimulation Versus Electro-acupuncture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for cardiovascular/respiratory disorder and geriaterics-faculty of physical therapy, Cairo University
Other Study IDs: P.T.REC/012/002523
Record Dates: First submitted 2019-12-20; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Salivation
MeSH Terms: conditions — Sialorrhea | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TENS group: Volunteers in this group (n=50) will receive only one session of 5-minute extra-oral TENS applied on bilateral parotid gland with 50 HZ frequency and pulse duration 250 µs.
  Interventions: Device: TENS
- electro-acupuncture group: Volunteers in this group (n=50) will receive only one session of 5-minute electro-acupuncture on local acu-points St4 and St 7 bilateraly with 2 HZ frequency.
  Interventions: Device: electro-acupuncture

INTERVENTIONS:
Device: TENS — Volunteers in this group (n=50) will receive only one session of 5-minute extra-oral TENS applied on bilateral parotid gland with 50 HZ frequency and pulse duration 250 µs.
  Groups: TENS group
Device: electro-acupuncture — Volunteers in this group (n=50) will receive only one session of 5-minute electro-acupuncture on local acu-points St4 and St 7 bilateraly with 2 HZ frequency.
  Groups: electro-acupuncture group

SUMMARY:
Between available therapies for dry mouth is electrostimulation. Using an extra-oral device like TENS - which result in a statistically significant - increases the quantity of whole salivary flow rate production in xerostomia patients. The use of acupuncture as an alternative treatment modality for xerostomia has been documented in the Western medical field since the 1980s. Observational studies have demonstrated that acupuncture treatment may increase salivary flow in healthy volunteers.

DETAILED DESCRIPTION:
It is possible that an increase of the blood fiux in the salivary glands may be one of the mechanisms behind the positive effect of acupuncture on the metabolism of the salivary glands, which leads to an increase of the salivary fiow.

Transcutaneous electric nerve stimulation (TENS) is a non-pharmacological and well known physical therapy modality which is widely for the acute and chronic pain management.

Electrostimulation using an extraoral device like TENS on parotid gland results in a statistically significant increase in the quantity of whole saliva flow rate production.

Starting a prevention program as early as possible considering the most practical, cost effective and efficient treatments with the best risk-benefit ratio will help to diminish dry mouth symptoms and sequelae.

ELIGIBILITY:
Inclusion Criteria:

- 1) 100 healthy adult volunteers from both sexes. 2) Application time of TENS and electro-acupuncture will be fixed for all volunteers between 9:00 am to 11:00 am.

3) The volunteers will be advised to have nothing to eat, drink, chew gum, coffee intake and oral hygiene before the test at least by one hour

Exclusion Criteria:

* 1) Volunteers under 18 years of age. 2) Pregnant females. 3) Habits (mouth breathing, smoking, alcohol and drug abuse). 4) Cancer patients (patients on chemotherapy/immunotherapy and history of head and neck radiotherapy).

  5) Cardiac patients (cardiac pacemakers and defibrillators). 6) Patients wearing hearing aids. 7) Chronic inflammatory autoimmune disease such as Sjogren's syndrome (an autoimmune disease that induces exocrine dysfunction and abnormalities), other rheumatologic diseases (including: rheumatoid arthritis, Systemic lupus erythematosus, scleroderma, mixed connective tissue disease, etc), sarcoidosis, amyloidosis, Crohn's disease and ulcerative colitis.

  8) Acute oral inflammatory disorders, gingivostomatitis, tonsillitis and dehydration.

  9) Infectious diseases e.g (HIV/AIDS, HCV and Tuberculosis). 10) Patients undergoing the use of any drugs. 11) Patients with neurological disorders: stroke, parkinson's disease, epilepsy, Bell's palsy, Alzheimer's disease, Patients with cerebrovascular problems, patients with a history of aneurysm and patients with transient ischaemia.

  12) Salivary gland diseases and disorders: agenesis of the salivary glands, sialoadenitis and sialolithiasis. Patients with Salivary duct ligation, history of salivary gland pathology, salivary gland inflammation and parotid gland infection.

  13) Psychogenic diseases and conditions: stress, anxiety, nervousness, depression, schizophrenia and eating disorders ( bulimia).

  14) Endocrine diseases: hyperthyroidism, hypothyroidism, Cushing's syndrome and Addison's disease and systemic diseases like diabetes mellitus.

  15) Others: cystic fibrosis, hypertension, fibromyalgia, chronic fatigue syndrome, burning mouth syndrome, primary biliary cirrhosis, liver transplant candidates, renal diseases, renal dialysis, anemia and atrophic gastritis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity card
Study Population: 100 healthy volunteers above 18 years from both sexes randomly assigned to TENS or electro-acupuncture group.
  * (TENS group): Volunteers in this group (n=50) will receive only one session of 5-minute extra-oral TENS applied on bilateral parotid gland with 50 HZ frequency and pulse duration 250microsecons
  * (Electro-acupuncture group): Volunteers in this group (n=50) will receive only one session of 5-minute electro-acupuncture on local acu-points St4 and St 7 bilateraly with 2 HZ frequency.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
salivary flow rate | during the five-minute TENS session.
  It is estimated as follow:
  * By dividing whole resting salivary volume on five minute collection period , thus whole resting salivary flow rate (ml/minute) is obtained (baseline).
  * Dividing stimulated salivary volume - collected during TENS application - on five minute collection period, thus stimulated salivary flow rate (ml/minute) is obtained.
  * Assessing improvement is done by comparing stimulated with whole resting salivary flow rate. Any increase in salivary rate will be considered an improvement

CONTACTS AND LOCATIONS:
Overall Officials: ali ismail, lecturer, Principal Investigator — Lecturer PT for Cardiovascular / Respiratory Disorder and Geriatrics
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt